CLINICAL TRIAL: NCT06591416
Title: Minimally Invasive Surgical Technique with and Without Granulation Tissue Preservation Using a Combination of Β Tri-Calcium Phosphate and Hyaluronic Acid Gel
Brief Title: Minimally Invasive Surgical Technique in Management of Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, yomna Medhat Elsaka, Principle investigator, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIST
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-04

CONDITIONS: Periodontal Diseases
Keywords: Minimally invasive surgical technique; Granulation tissue preservation; infrabony defect
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minimally invasive surgical technique with total removal of granulation tissue (Active Comparator): Minimally invasive surgical technique with total removal of granulation tissue
  Interventions: Procedure: minimally invasive surgical technique
- Minimally invasive surgical technique with partial removal of granulation tissue (Experimental): Minimally invasive surgical technique with partial removal of granulation tissue
  Interventions: Procedure: minimally invasive surgical technique with granulation tissue preservation

INTERVENTIONS:
Procedure: minimally invasive surgical technique — minimally invasive surgical technique
  Arms: Minimally invasive surgical technique with total removal of granulation tissue
Procedure: minimally invasive surgical technique with granulation tissue preservation — minimally invasive surgical technique with granulation tissue preservation
  Arms: Minimally invasive surgical technique with partial removal of granulation tissue

SUMMARY:
In the fast-growing era of contemporary periodontology, the understanding of biological concepts in wound healing together with the evolution of the flap design and biomaterials applied in periodontal regeneration allowed for improved minimally invasive surgical techniques. As minimally invasive approaches reduce the surgical trauma, maintain soft tissue support which allow stable primary closure of the wound. These advantages have led more researchers to apply the concept of minimally invasive surgical techniques (MISTs) in the treatment of infrabony lesions.

Granulation tissue is an immature connective tissue that appears naturally during chronic inflammation or wound healing. This tissue is not a cause of periodontitis.

So, no need to remove it during periodontal treatment. The aim of preservation of the defect-filling granulation tissue after detachment of its base is assumed to act as a soft tissue support, and to increase wound stability especially in the area of the interdental papilla and avoid post-operative marginal recession. One of the alloplastic bone grafts is βeta tri-calcium phosphate (β-TCP). β-TCP has been widely used in periodontal regeneration, where many studies used beta tri-calcium phosphate alone or in combination with other grafting materials in different surgical regenerative procedures have shown promising results for bone filling and new vital bone formation. Hyaluronic acid gel shows anti-inflammatory, antibacterial, and antioxidant properties in the treatment of periodontal diseases. In addition, due to its viscoelastic properties, it can be used as an adjunct to maintain space during periodontal tissue regeneration.

A concentration of 0.8% hyaluronic acid gel has been used effectively in the non-surgical and surgical management of periodontal diseases.

Aim of The Study The aim of the present study is to evaluate the effects of the minimally invasive surgical technique with and without granulation tissue preservation using a combination of beta tri calcium phosphate and hyaluronic acid gel.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ranged from 30 to 50 years old for both genders.
2. Patients are medically free according to the American society of anesthesiologists (ASA) considered as ASA I.
3. The selected participants with a diagnosis stage III grade B periodontitis.
4. Defect morphology: Isolated interproximal infrabony defect of at least 5mm CAL which does not extend beyond the adjacent interproximal region.
5. Optimal compliance as assessed during the case related phase I therapy and evidenced by no missed treatment appointments and positive attitude toward oral hygiene.
6. Bleeding on probing <25%.

Exclusion Criteria:

1. Smoker and pregnant patients.
2. Multiple, interconnected vertical defects.
3. Generalized horizontal bone defects.
4. Teeth with incorrect endodontic treatment or restoration.
5. Stage I, II or IV periodontitis.
6. Patient who need complex prosthetic rehabilitation.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level | 6 months
  measured from cemento-enamel junction to the base of the pocket by using william's graduated periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Gharbia Governement, Egypt

IPD SHARING:
Plan to Share IPD: No